CLINICAL TRIAL: NCT00367783
Title: A 12-Week, Phase 2A, Randomized, Subject And Investigator Blind, Placebo-Controlled Trial To Evaluate The Effect Of CP-741,952 On Weight Loss In Otherwise Healthy Overweight And Obese Adult Subjects
Brief Title: Safety, Toleration and Efficacy of CP-741,952 for the Treatment of Obesity
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See Detailed Description for termination reason.
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A7081004
Record Dates: First submitted 2006-05-30; First posted 2006-08-23 (Estimated); Last update posted 2011-08-01 (Estimated); Status verified 2011-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CP-741,952

SUMMARY:
The purpose of this study is to determine whether CP-741,952 is effective in the treatment of obesity and to determine 12 week safety and toleration.

DETAILED DESCRIPTION:
Following review of the preliminary data from completed study A7081004, the development program for CP-741,952 was terminated on 15 March 2007. Primary reasons for program termination included a lack of significant efficacy at all doses investigated and an increased incidence of mild to moderate elevations in serum transaminases, primarily alanine aminotransferase (ALT), and liver fat content, in treated compared to placebo subjects. A synopsis will be created and will include greater detail on these findings.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 30-40 kg/m2

Exclusion Criteria:

* Women of childbearing potential

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-06; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Weight Loss, toleration, safety

SECONDARY OUTCOMES:
Waist Circumference, serum lipids

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Kalamazoo, Michigan
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, San Antonio, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7081004&StudyName=Safety%2C%20Toleration%20and%20Efficacy%20of%20CP-741%2C952%20for%20the%20Treatment%20of%20Obesity